CLINICAL TRIAL: NCT06924333
Title: The Skin Microbiota in Skin Disease and Eczema
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-06196-02
Record Dates: First submitted 2025-01-27; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Skin Disease; Eczema; Eczema Atopic Dermatitis
MeSH Terms: conditions — Skin Diseases; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin microbiota, skin specimens, blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with atopic eczema, eczema or other skin diseases

SUMMARY:
Background: The skin microbiota influence skin health in several skin diseases and atopic dermatitis (AD). Presence of Staphylococcus have been associated to a sever course of the disease.

Objectives: The aim of the study is to investigate the influence of bacteria, and the skin microbiota on the inflammation and skin barrier. Moreover, dysbiosis in the microbiota, the inflammation profile, the skin barrier damage will be related to objective and patient oriented measures.

Importance: Knowledge of interactions between host defense, skin barrier and bacterial colonizing skin can facilitate development of new prevention and treatment strategies to control microbial impact in skin diseases and eczema.

DETAILED DESCRIPTION:
The role of the skin microbiome in atopic eczema and other skin diseases remains to be investigated. There are reports indicating an association of skin-colonization of Staphylococcus aureus (S. aureus) and the severity of the disease. Skin colonizing pathogens might be important cofactor for persistence of eczema and other skin diseases, as well as the commensal, non-pathogenic, microflora of the skin might have protective effects. The aim of this research project is to investigate the skin microbiome in patients with eczema and other skin diseases and elucidate the relation to skin barrier impairment and severity of the skin disease.

Specifically, we will:

* Determine the skin microbiome and metagenome in skin of patients with eczema and other skin diseases.
* Straighten out the relationship between the skin microbiome, the skin barrier, contact allergies, quality of life, eczema control and severity in patients with eczema and other skin diseases.
* Identify biological markers, such as antimicrobial peptides, cytokines and gene-expression profiles in skin, and other factors contributing to the development and persistence of eczema and other skin diseases.

ELIGIBILITY:
Inclusion Criteria: Skin diseas, atopic eczema, eczema

-

Exclusion Criteria:

* Inabillity to give informed concent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patints with skin diseases, atopic eczema and eczema. Healthy volonteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Skin microbiota | At baseline/enrollment through study completion, an average of 1 year.
  Characterization of skin microbiota are assessed at skin of patients with eczema or skin disease.
Skin Barrier impairment tewl | At baseline/enrollment through study completion, an average of 1 year.
  meassurment of trans epidermal water loss (g/m2h)
EASI | At baseline/enrollment through study completion, an average of 1 year.
  Eczema area and severity index are assessed (score 0-72)
Patient oriented outcome measures RECAP | At baseline/enrollment through study completion, an average of 1 year.
  Recap of atopic eczema, RECAP. RECAP is a seven-item questionnaire designed to capture the experience of eczema control in all ages and eczema severities.
Patient oriented outcome measures POEM | At baseline/enrollment through study completion, an average of 1 year.
  The Patient Oriented Eczema Measure (POEM) is a tool used for monitoring atopic eczema severity. It focuses on the illness as experienced by the patient.
Patient oriented outcome measures DLQI | At baseline/enrollment through study completion, an average of 1 year.
  The DLQI is designed to measure the health-related quality of life of adult patients suffering from a skin disease.
Patient oriented outcome measures NRS Itch | At baseline/enrollment through study completion, an average of 1 year.
  The Peak Pruritus Numerical Rating Scale (NRS) is a well-defined, reliable, fit-for-purpose measure to evaluate patient-reported intensity of worst itch in the previous 24 h for adults with moderate-to-severe atopic dermatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
If confidential